CLINICAL TRIAL: NCT01862445
Title: A Retrospective Study to Assess the Efficacy and Safety of Chlorambucil Plus Rituximab as Front-line Therapy in Elderly and/or Unfit Patients Affected by B-cell Chronic Lymphocytic Leukemia
Brief Title: Retrospective Study: Efficacy and Safety of Chlorambucil + Rituximab in CLL Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: LLC1013
Record Dates: First submitted 2013-05-17; First posted 2013-05-24 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: CLL; B-cell; Small Lymphocytic Lymphoma; Untreated B-CLL; Elderly Patients
Keywords: Chronic Lymphoid Leukemia, Chlorambucil, Rituximab
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, B-Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study group: Patients receiving Chlorambucil plus Rituximab

SUMMARY:
This is a non interventional study to evaluate the efficacy and safety of Chlorambucil plus Rituximab as firstline therapy in elderly and/or unfit patients affected by B-cell Chronic Lymphocytic Leukemia (B-CLL).

DETAILED DESCRIPTION:
Illness: treatment overview Chronic lymphocytic leukemia (B-CLL) is the most prevalent adult leukemia among western countries (6.7% Non-Hodgkin Lymphomas- NHL). The incidence rate is 2-6 cases per 100.000 person per year increasing with age and reaching an incidence rate of about 13/100.000 at 65 years, median age of onset of the disease. There are two clinical staging systems currently in use for CLL (Rai and Binet staging systems) allowing a rough division of patients into three prognostic groups: good, intermediate and poor prognosis. The clinical course ranges from an indolent behaviour (Rai 0, Binet A) with a long term survival to an aggressive disease with a median survival of 2 years (Rai III and IV, Binet C). There is non survival benefit associated with an early therapy (Binet stage A and B). Treatment usually is initiated when patient progress to the advanced stage (Binet stage C) and/or become symptomatic (fever, night sweats, weight loss). Purine-analogues based chemo-immunotherapy regimens are now considered the standard of care for fit patient with B-CLL (Fludarabine-Cyclophosphamyde-Rituximab, FCR regimen). But aging of the host and biological features of the disease are critical issues in the choice of therapy. The FCR regimen can result in significant myelosuppression and a high rate of early and late infections, especially in elderly patients with B-CLL, suggesting that it may be too toxic and therefore unsuitable for the large subpopulation of elderly and comorbid patients affected by B-CLL/SLL.

Rationale Chlorambucil, an alkylating agent, was the standard first line treatment for B-CLL/SLL before the development of the purine analogues and monoclonal antibodies. Later, phase III trials showed an improved ORR and a prolongation of PFS with fludarabine alone. A further improvement was obtained with the addition of Cyclophosphamide to Fludarabine. Eventually, Fludarabine in combination with Cyclophosphamide and the monoclonal anti-CD20 antibody Rituximab became the standard first line therapy for CLL patients 18 to 65 years old. At the same time, the FCR regimen showed a significant rate of early toxicity consisting of myelosuppression and infection and also a high rate of late infection. Data showed by Hallek et al reported a rate of grade 3-4 hematological toxicity and total infections of 56% and 25%, respectively. They reported 8 treatment-related deaths (2%), five of these due to infections and 4 deaths occurring before the 3th cycle. Also has been reported by Tam et al a risk of 10% of late infection for the first year of remission after FCR treatment. Low-dose FCR was evaluated as an alternative option showing a lower rate of neutropenia, without reduction of response rate. Nevertheless, it was demonstrated to reduce the PFS and it has not been evaluated in the elderly or medically unfit population. Alternative treatments (i.e., low-dose fludarabine, low-dose fludarabine plus cyclophosphamide, rituximab alone) have been explored in phase II trials in elderly and/or medically unfit patients with CLL. Since the cohort sizes were small, however, no definitive recommendations could be made for clinical practice. About three-quarters of CLL patients are more than 65 years old. Data from the CLL 5 phase III trial of GCLLSG (German CLL study group) comparing fludarabine vs Chlorambucil in this setting of patients (median age 70 years, range 65-80 years) displayed no differences in OS and PFR between Fludarabine and Chl, despite a greater percentage of CR and ORR with Fludarabine. This suggests that in elderly B-CLL patients, Fludarabine alone does not represent a major benefit in respect of Chl as front-line therapy. However, rates of complete response (CR) with front-line Chlorambucil single agent are relatively low (up to 7%) as are overall responses (approximately 65%). Phase II trials are ongoing to investigate the efficacy and safety of Rituximab in combination with Chl in previously untreated patients affected by B-CLL.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of B-CLL or Small Lymphocytic Lymphoma (SLL) according to the World Health Organisation (WHO) classification 2008;
* Previously untreated B-CLL requiring therapy according to the NCI criteria (Hallek M et al, Blood 2008 (Appendix G) undergone to first line of therapy with Chl-R;
* All patients included in the study must have started treatment by December 2011;
* Age ≥ 65 years or unfit pts ≥ 18 years old with a CIRS score ≥7 (Appendix E);
* Eastern Cooperative Oncology Group Performance Status Grade of 0-2 (Appendix B) ;
* Life expectancy > 6 months;
* Signed written informed consent according to ICH/EU/GCP and national local law.

Exclusion Criteria:

* Patients who have received prior therapy: chemotherapy and/or immunotherapy, stem cell transplantation, investigational drugs administered to treat B-CLL before Chl-R;
* Transformation of B-CLL to aggressive lymphomas (Richter's Syndrome);
* One or more individual organ/system impairment score of 4 as assessed by CIRS definition;
* HIV infection;
* Active, uncontrolled HCV and/or HBV infections or liver cirrhosis;
* Patients who started Chl-R after December 2011.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The GIMEMA Chronic Lymphocytic Leukemia Working Party promotes an observational, retrospective, multicenter study on safety and efficacy of Chl-R administered front-line to treat elderly and/or unfit pts affected by B-CLL.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-10; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Number of responding patients. | 10 months from study entry
  Overall response rate.

SECONDARY OUTCOMES:
Number of adverse events. | 24 months from study entry
  Safety of Rituximab and Chlorambucil regimen (type, frequency and severity).
Number of days from the first dose of treatment to re-treatment. | 24 months from study entry.
  Time to Re-Treatment (TTR) estimation starting from the date of the first dose of the study drug
Number of patients surviving. | 24 months from study entry.
  Progression Free Survival (PFS) estimation starting from the date of the first dose of the study drug.
  Overall Survival (OS) estimation starting from the date of the first dose of the study drug
Number of patients in which the response and the biological and clinical characteristics of the disease at baseline are associated. | After 10 months from study entry.
  Fitness status, FISH, IgVH, Zap70 and CD38.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Laurenti, Dr., Study Chair — Istituto di Ematologia, Università Cattolica del Sacro Cuore di Roma
Locations (20):
- Italy (20):
  - U.O.C. Ematologia e Terapia Cellulare - Ospedale "C. e G. Mazzoni" di Ascoli Piceno, Ascoli Piceno
  - UOC Ematologia Ospedale " Monsignor Raffaele Dimiccoli", Barletta
  - Azienda Ospedaliera Pugliese Ciaccio - Presidio Ospedaliero A.Pugliese - Unità Operativa di Ematologia, Catanzaro
  - Sezione di Ematologia e Fisiopatologia delle Emostasi, Ferrara
  - Policlinico di Careggi, Florence
  - Struttura Complessa di Ematologia Ospedali Riuniti Foggia - Azienda Ospedaliero-Universitaria, Foggia
  - Divisione di Ematologia - Azienda Ospedaliera Ospedali Riuniti "Papardo Piemonte", Messina
  - UO Ematologia - AOU Policlinico di Modena, Modena
  - U.O. di Oncoematologia di Nocera Inferiore-plesso ospedaliero "A. Tortora" di Pagani del DEA Nocera-Pagani, Nocera Inferiore
  - Cattedra di Ematologia CTMO Università degli Studi di Parma, Parma
  - Div. di Ematologia di Muraglia - CTMO Ospedale San Salvatore, Pesaro
  - Dipartimento Emato-Oncologia A.O."Bianchi-Melacrino-Morelli", Reggio Calabria
  - U.O. di Ematologia - Centro Oncologico Basilicata, Rionero in Vulture
  - U.O.C. Ematologia - Ospedale S.Eugenio, Roma
  - U.O.S.A. Ematologia ASL RMA Presidio Nuovo Regina Margherita, Roma
  - Università Cattolica del Sacro Cuore - Policlinico A. Gemelli, Roma
  - Università degli studi "Sapienza" di Roma, Roma
  - A.O. Santa Maria - Terni S.C Oncoematologia, Terni
  - Divisione di Ematologia dell' Università degli Studi di Torino - "Città della Salute e della Scienza di Torino", Torino
  - Struttura Complessa II Medicina - Ematologia - Centro di Riferimento Ematologico - Ospedale Maggiore, Trieste

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: GIMEMA Foundation website — http://www.gimema.it